CLINICAL TRIAL: NCT03890328
Title: Radiofrequency-assisted Splenic Preservation Versus Conventional Treatment of Blunt Splenic Injury: A Prospective Cohort Study.
Brief Title: RF-assisted Splenic Preservation VS Conventional Treatment of Blunt Splenic Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Hospital, China (Other)
Collaborators: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, fengkai, associate professor, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81672857
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2009-03

CONDITIONS: Radiofrequency Can be Used to Treat Splenic Trauma Because of Its Excellent Coagulation Hemostasis
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RF group (Experimental): radiofrequency-assisted spleen-preserving therapy group.
  Interventions: Procedure: radiofrequency ablation
- CT group (No Intervention): Conventional Treatment of Blunt Splenic Injury group.

INTERVENTIONS:
Procedure: radiofrequency ablation — apply RF therapy to the treatment of splenic trauma
  Arms: RF group

SUMMARY:
Radiofrequency (RF) can be used to treat splenic trauma because of its excellent coagulation hemostasis. This study aimed to compare the efficacy of RF-assisted spleen-preserving surgery with that of conventional splenorrhaphy/splenectomy in the treatment of blunt splenic injury.

A total of 122 patients with splenic trauma admitted to two tertiary referral centers from June 2011 to June 2014 were included in this prospective cohort study. The 67 patients at one center were treated by radiofrequency-assisted spleen-preserving therapy (RF group), and the 55 patients admitted at the other center underwent conventional treatment (CT group). Demographics and clinical characteristics of the two groups were comparable.

Compared to traditional splenorrhaphy and splenectomy, RF-assisted splenic hemostasis and salvage was safe, effective and easy to use in the treatment of splenic injuries. In particular for high-grade splenic injuries, these techniques preserved sufficient splenic tissue without any increase in patients with surgical risk.

ELIGIBILITY:
Inclusion Criteria：

1. age below 70
2. blunt abdominal injury combined with indication of post-traumatic splenectomy according to the guidelines provided by the Society for Surgery of the Alimentary Tract in 2005
3. patients transferred directly to the trauma center after injury who had not been treated by any specific spleen-directed therapy in the transferring hospital
4. AAST grade II splenic injury with hemodynamic instability or progressive bleeding requiring active intervention
5. AAST grade Ⅲ-Ⅳsplenic injury, or splenic laceration involving less than 50% of the splenic parenchyma

Exclusion Criteria:

1. penetrating abdominal injury
2. concomitant organ injury with an abbreviated injury scale (AIS) greater than 4 that threatened the life of the patient
3. excessive vascular injury to the splenic pedicle or substantial devitalized splenic tissues when it was expected in when less than 25% of the spleen could be preserved
4. patients who had failed NOM
5. patients with pathologic splenic rupture

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
Mean operative time， | intraoperative
  Mean operative time of the RF group was compared with that of CT group.
intraoperative bleeding | intraoperative
  Intraoperative bleeding of the RF group was compared with that of CT group.

CONTACTS AND LOCATIONS:
Overall Officials: Kuansheng Ma, Ph.D, Principal Investigator — Institute of hepatobiliary surgery,Southwest Hospital
Locations (1):
- Institute of hepatobiliary surgery,Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No